CLINICAL TRIAL: NCT00133133
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Analgesic Efficacy, Safety and Tolerability of ALGRX 4975 in Subjects After Open Cholecystectomy
Brief Title: Efficacy and Safety of ALGRX 4975 in the Treatment of Postoperative Pain After Gall Bladder Removal
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AlgoRx Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4975-2-011-2
Record Dates: First submitted 2005-08-18; First posted 2005-08-22 (Estimated); Last update posted 2006-12-20 (Estimated); Status verified 2006-02

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Open cholecystectomy; Capsaicin
MeSH Terms: conditions — Pain, Postoperative

INTERVENTIONS:
Drug: ALGRX 4975

SUMMARY:
Postoperative pain after gall bladder removal can be significant, mobility limiting and extend hospital stay. ALGRX 4975 is an ultra-pure form of capsaicin, which is a pain medicine that has the potential for long-term pain relief following a single administration. This study will determine whether ALGRX 4975 can provide pain relief following gall bladder removal.

DETAILED DESCRIPTION:
Postoperative pain after open cholecystectomy can be significant and mobility limiting, causing increased risk of deep venous thrombosis, pulmonary complications, and extended hospital stay. With increasing emphasis on early postoperative mobilization, adequate postoperative pain control is essential. Acute postoperative pain is currently managed largely with opioids and co-administration of nonsteroidal anti-inflammatory drugs (NSAIDS). Opioids are highly effective in managing acute postoperative pain, however dosing is often limited by side effects such as respiratory depression, nausea and vomiting, and sedation. NSAIDS are administered to reduce opioid use, but may also have limiting side effects, such as gastrointestinal toxicity and platelet dysfunction. New strategies to manage acute postoperative pain would provide clinical benefit. ALGRX 4975 is an ultra-pure form of capsaicin, which is a pain medicine that has the potential for long-term pain relief following a single administration. This study will determine whether ALGRX 4975 can provide pain relief following open cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing open cholecystectomy with the subcostal approach for cholelithiasis/cholecystitis
* American Society of Anesthesiologists (ASA) Class I or II

Exclusion Criteria:

* Active pancreatitis, any obstruction of the biliary tree, or hyperbilirubinemia (total bilirubin > 2.5 mg/dL)
* Previous abdominal surgical procedure with the exception of inguinal hernia repair or appendectomy by the lateral approach or cesarean section or hysterectomy if the surgery was performed more than 1 year prior to study participation and the subject experienced no postoperative complications
* Diabetes mellitus with HbA1C > 9.5 or a history of prolonged uncontrolled diabetes mellitus
* Systolic blood pressure greater than 150 mmHg or diastolic greater than 95 mmHg

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2005-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Average numeric rating scale (NRS) scores for pain on ambulation assessed in the evening on the day of surgery and the first four postoperative days

SECONDARY OUTCOMES:
Time to first use and total supplemental pain medication use
NRS scores for pain on the first 14 days postoperatively
Spirometry on postoperative days 1 to 4
Safety and tolerability
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Slobodan Krstic, MD, Principal Investigator — Emergency Center, Clinical Center of Serbia
Locations (1):
- Emergency Center, Clinical Center of Serbia, Belgrade, Serbia and Montenegro